CLINICAL TRIAL: NCT01438996
Title: A Phase 2, Open-label, Single-center, Extension Study to Evaluate the Booster Response Induced by Vi-CRM197 After Priming With Either Vi-CRM197 or Typherix Administered in Adult Subjects in H01_04TP Study (NCT01193907)
Brief Title: Extension Study of H01_04TP to Evaluate the Booster Response Induced by Vi-CRM197 in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H01_04E1TP
Record Dates: First submitted 2011-09-19; First posted 2011-09-22 (Estimated); Results first posted 2014-03-24 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-02

CONDITIONS: Typhoid Fever
Keywords: Typhoid fever; Glycoconjugate vaccine; Vi polysaccharide; Immunogenicity
MeSH Terms: conditions — Typhoid Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- NVGH Vi-CRM/NVGH Vi-CRM (Experimental): One 0.5 mL dose of NVGH Vi-CRM197 5.0 mcg in adults who received 1 dose of NVGH Vi-CRM197 5.0 mcg in H01_04TP study
  Interventions: Biological: NVGH Vi-CRM197
- Vi-PS/NVGH Vi-CRM (Experimental): One 0.5 mL dose of NVGH Vi-CRM197 5.0 mcg in adults who received 1 dose of Vi-polysaccharide (PS) in H01_04TP study
  Interventions: Biological: NVGH Vi-CRM197
- NVGH Vi-CRM (Experimental): One 0.5 mL dose of NVGH Vi-CRM197 5.0 mcg in naive adults
  Interventions: Biological: NVGH Vi-CRM197

INTERVENTIONS:
Biological: NVGH Vi-CRM197 — Vi-CRM197 glycoconjugated vaccine

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and the kinetics of the anti-Vi antibody response following secondary vaccination with the Novartis Vaccines Institute for Global Health (NVGH) Vi-CRM197 vaccine in healthy adults previously vaccinated with either the NVGH Vi-CRM197 or Vi-polysaccharide (Typherix) in the H01_04TP study (NCT01193907) and the immunogenicity and the kinetics of the anti-Vi antibody response following primary vaccination with the NVGH Vi-CRM197 vaccine in naïve healthy adults.

ELIGIBILITY:
Inclusion criteria

All Subjects:

1. Males and females of age ≥18 to ≤42 years.
2. Individuals, who, after the nature of the study have been explained to them, have given written consent according to local regulatory requirements.
3. Individuals in good health as determined by the outcome of medical history, physical examination and clinical judgment of the investigator.
4. If women, use of birth control one month before study start, a negative pregnancy test and willingness to use birth control measures for the entire study duration.

   H01_04TP subjects only:
5. Individuals who previously participated in the H01_04TP study and were vaccinated with either NVGH Vi-CRM197 (5μg) or with the licensed Vi-PS.
6. Individuals who have received no Vi vaccination subsequent to the one received in the H01_04TP study.

Inclusion criteria

All subjects:

1. Individuals with behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the subject's ability to participate in the study.
2. Individuals with any progressive or severe neurological disorder, seizure disorder or Guillain-Barré syndrome.
3. Individuals who are not able to understand and to follow all required study procedures for the whole period of the study.
4. Individuals with history of any illness that, in the opinion of the investigator, pose additional risk to the subjects due to participation in the study.
5. Individuals with known or suspected HIV infection or HIV related disease, with history of an autoimmune disorder or any other known or suspected impairment /alteration of the immune system, or under immunosuppressive therapy including use of systemic corticosteroids or chronic use of inhaled high-potency corticosteroids within the previous 30 days, or were in chemotherapy treatment within the past 6 months.
6. Individuals with a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
7. Individuals with any serious chronic or progressive disease according to judgment of the investigator (e.g., neoplasm, insulin dependent diabetes, cardiac, renal or hepatic disease).
8. Individuals who have any malignancy or lymphoproliferative disorder.
9. Individuals with history of allergy to vaccine components.
10. Individuals participating in any clinical trial with another investigational product 30 days prior to first study visit or intent to participate in another clinical study at any time during the conduct of this study.
11. Individuals who received any vaccines within 4 weeks prior to enrolment in this study or who are planning to receive any vaccine within 4 weeks from the study vaccine
12. Individuals who have received blood, blood products and/or plasma derivatives including parenteral immunoglobulin preparations in the past 12 weeks.
13. Individuals who are part of study personnel or close family members to the personnel conducting this study.
14. Individuals with body temperature > 38.0 degrees Celsius within 3 days of intended study immunization.
15. BMI > 35 kg/m2.
16. Individuals with history of substance or alcohol abuse within the past 2 years.
17. Women who are pregnant or breast-feeding or of childbearing age who have not used any birth control measure one month prior to study start or do not plan to use acceptable birth control measures, for the duration of the study.
18. Females with history of stillbirth, neonatal loss, or previous infant with anomaly.
19. Individuals who have a previously ascertained or suspected disease caused by S. Typhi.
20. Individuals who have had household contact with/and or intimate exposure to an individual with laboratory confirmed S. Typhi.
21. Any condition which, in the opinion of the investigator may interfere with the evaluation of the study objectives.

    Naïve subjects only:
22. Individuals who have previously received any vaccine against typhoid fever (either oral live attenuated or injectable vaccines)

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Van Damme, MD, Principal Investigator — Universiteit Antwerpen
Locations (1):
- Centre for the Evaluation of Vaccination (CEV), Antwerp, Wilrijk, Belgium

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled: 17 OCT 11, Last subject completed: 13 DEC 11.
Period: Overall Study
Arm/Group | NVGH Vi-CRM/NVGH Vi-CRM | Vi-PS/NVGH Vi-CRM | NVGH Vi-CRM
Started | 18 | 13 | 20
Completed | 14 | 12 | 20
Not Completed | 4 | 1 | 0
Not completed — Not meeting Inclusion Criteria | 4 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NVGH Vi-CRM/NVGH Vi-CRM | Vi-PS/NVGH Vi-CRM | NVGH Vi-CRM | Total
Number analyzed (Participants) | 18 | 13 | 20 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 13 | 20 | 51
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (5.8) | 26.3 (6.6) | 26.0 (6.2) | 25.8 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 10 | 17
  Male | 13 | 11 | 10 | 34
Region of Enrollment [Number; unit: participants]
  Belgium | 18 | 13 | 20 | 51

OUTCOME MEASURES:

1. Primary Outcome: Anti-Vi ELISA Geometric Mean Concentration (GMC)
Description: To evaluate the immunogenicity and the kinetics of the immune response induced by one dose of NVGH Vi-CRM197 at study day 3 after vaccination as as measured by enzyme-linked immunosorbent assay (ELISA)
Time Frame: At 3 days after vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA Units/mL
Arm/Group | NVGH Vi-CRM/NVGH Vi-CRM | Vi-PS/NVGH Vi-CRM | NVGH Vi-CRM
Number analyzed (Participants) | 14 | 12 | 20
ELISA Units/mL | 35 [18 to 65] | 31 [16 to 60] | 3.22 [1.99 to 5.23]

2. Primary Outcome: Anti-Vi ELISA GMC
Description: To evaluate the immunogenicity and the kinetics of the immune response induced by one dose of NVGH Vi-CRM197 at study day 7 after vaccination as as measured by ELISA
Time Frame: At 7 days after vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA Units/mL
Arm/Group | NVGH Vi-CRM/NVGH Vi-CRM | Vi-PS/NVGH Vi-CRM | NVGH Vi-CRM
Number analyzed (Participants) | 14 | 12 | 20
ELISA Units/mL | 65 [42 to 102] | 40 [24 to 67] | 20 [10 to 39]

3. Primary Outcome: Anti-Vi ELISA GMC
Description: To evaluate the immunogenicity and the kinetics of the immune response induced by one dose of NVGH Vi-CRM197 at study day 28 after vaccination as as measured by ELISA
Time Frame: At 28 days after vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA Units/mL
Arm/Group | NVGH Vi-CRM/NVGH Vi-CRM | Vi-PS/NVGH Vi-CRM | NVGH Vi-CRM
Number analyzed (Participants) | 14 | 12 | 20
ELISA Units/mL | 44 [28 to 69] | 50 [35 to 71] | 111 [78 to 156]

4. Primary Outcome: Percentage of Subjects With at Least 4-fold Increase in Anti-Vi ELISA Titers
Time Frame: At 3 days after vaccination as compared to baseline
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | NVGH Vi-CRM/NVGH Vi-CRM | Vi-PS/NVGH Vi-CRM | NVGH Vi-CRM
Number analyzed (Participants) | 14 | 12 | 20
percentage of subjects | 0 [0 to 23] | 0 [0 to 26] | 0 [0 to 17]

5. Primary Outcome: Percentage of Subjects With at Least 4-fold Increase in Anti-Vi ELISA Titers
Time Frame: At 7 days after vaccination as compared to baseline
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | NVGH Vi-CRM/NVGH Vi-CRM | Vi-PS/NVGH Vi-CRM | NVGH Vi-CRM
Number analyzed (Participants) | 14 | 12 | 20
percentage of subjects | 7 [0 to 34] | 0 [0 to 26] | 60 [36 to 81]

6. Primary Outcome: Percentage of Subjects With at Least 4-fold Increase in Anti-Vi ELISA Titers
Time Frame: At 28 days after vaccination as compared to baseline
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | NVGH Vi-CRM/NVGH Vi-CRM | Vi-PS/NVGH Vi-CRM | NVGH Vi-CRM
Number analyzed (Participants) | 14 | 12 | 20
percentage of subjects | 0 [0 to 23] | 17 [2 to 48] | 100 [83 to 100]

7. Secondary Outcome: Number of Subjects Reporting Any (Local, Systemic and Other) Post Vaccination Reaction
Description: Solicited reactions collected during the 7-day period after vaccination are pain, erythema, induration, chills, malaise, myalgia, headache, arthralgia, fatigue and fever.
Time Frame: During the 7-day period after vaccination
Measure: Number; unit: participants
Arm/Group | NVGH Vi-CRM/NVGH Vi-CRM | Vi-PS/NVGH Vi-CRM | NVGH Vi-CRM
Number analyzed (Participants) | 14 | 12 | 20
participants | 14 | 12 | 18

8. Secondary Outcome: Number of Subjects Reporting AE
Description: AE during 28 days after vaccination(including solicited reactions during 7 days after vaccination)
Time Frame: During the 28-day period after vaccination
Measure: Number; unit: participants
Arm/Group | NVGH Vi-CRM/NVGH Vi-CRM | Vi-PS/NVGH Vi-CRM | NVGH Vi-CRM
Number analyzed (Participants) | 14 | 12 | 20
participants | 14 | 12 | 20

9. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Time Frame: During the 28-day period after vaccination
Measure: Number; unit: participants
Arm/Group | NVGH Vi-CRM/NVGH Vi-CRM | Vi-PS/NVGH Vi-CRM | NVGH Vi-CRM
Number analyzed (Participants) | 14 | 12 | 20
participants | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | NVGH Vi-CRM/NVGH Vi-CRM | Vi-PS/NVGH Vi-CRM | NVGH Vi-CRM
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/12 | 0/20
Other Adverse Events (participants affected / at risk) | 14/14 | 12/12 | 20/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NVGH Vi-CRM/NVGH Vi-CRM (N=14) | Vi-PS/NVGH Vi-CRM (N=12) | NVGH Vi-CRM (N=20)
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1
diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
nausea (Gastrointestinal disorders) | 1 | 1 | 0
chills (General disorders) | 3 | 1 | 1
fatigue (General disorders) | 7 | 7 | 5
injection site erythema (General disorders) | 3 | 0 | 0
injection site induration (General disorders) | 0 | 0 | 4
injection site pain (General disorders) | 14 | 10 | 15
malaise (General disorders) | 4 | 6 | 5
gastroenteritis (Infections and infestations) | 1 | 1 | 1
nasopharingitis (Infections and infestations) | 6 | 3 | 3
oral herpes (Infections and infestations) | 0 | 1 | 1
rhinitis (Infections and infestations) | 2 | 0 | 0
arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
myalgia (Musculoskeletal and connective tissue disorders) | 4 | 2 | 2
dizziness (Nervous system disorders) | 1 | 0 | 0
headache (Nervous system disorders) | 6 | 8 | 9
syncope (Nervous system disorders) | 1 | 0 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event that no publication of the Study results has been made by NVGH within twelve (12) months of Study database lock and no proposed publication is under discussion by the publication committee, Principal Investigator may publish its own Study results, provided that he furnishes NVGH with a copy of the proposed publication for NVGH's review and comment, at least 1 month prior to submission to a publisher or disclosure to any third party.